CLINICAL TRIAL: NCT06698341
Title: UNdeRstAnding Novel Variants in AcutE MyocardiaL Infarction in Young Adults
Acronym: UNRAVEL
Status: Recruiting | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/00687
Record Dates: First submitted 2024-10-28; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-01

CONDITIONS: Myocardial Infarction, Acute
MeSH Terms: conditions — Myocardial Infarction | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 3X 6mL K2-EDTA tubes, 1X 3mL K2-EDTA tubes and 1X 3.5mL SST tube will be collected per subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Age ≤50 years old irrespective of the presence of CV risk factors* at the time of myocardial infarction
  Interventions: Procedure: Blood Draw
- Group 2: Age 51-60 years old with no more than 2 CV risk factor at the time of myocardial infarction, excluding diabetes mellitus
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw — 3X 6mL K2-EDTA tubes, 1X 3mL K2-EDTA tubes and 1X 3.5mL SST tube - 24.5ml of blood will be collected from patient

SUMMARY:
Cardiovascular disease (CVD) imposes significant mortality and morbidity worldwide. However, large gaps in our knowledge of CVD still exist. The clinical conundrum of the extremes of spectrums of CVD continues to baffle clinicians and researchers alike. These include patients without any major cardiovascular (CV) risk factors developing acute myocardial infarction (AMI) at a relatively young age (<50-60 years old), while at the other end of the spectrum, there are also patients with multiple CV risk factors but with minor or no coronary artery disease. These suggest the presence of other factors that predispose these patients to AMI.Recent advancements in technology, especially in the field of genomics, metabolomics, and proteomics, have led to exciting developments in our understanding of the development and prevention of CVD and AMI. In this study, the investigators aim to identify novel gene variants associated with the onset of MI in relatively young patients with minimal standard CV risk factors such as diabetes, obesity, hypertension and hypercholesterolaemia.Through genomic, metabolomics and proteomics analyses, this may better improve our understanding of the development of CVD and AMI, potentially developing novel preventive measures to reduce the risk or delay the onset as well as tailoring management plans to improve treatment outcomes and reduce adverse events for the patients.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) imposes significant mortality and morbidity worldwide. Large population-based studies in Western cohorts have formed the foundations of our knowledge on the traditional risk factors of cardiovascular disease. Despite this, large gaps in our knowledge of CVD still exist. The clinical conundrum of the extremes of spectrums of CVD continues to baffle clinicians and researchers alike. These include patients without any major cardiovascular (CV) risk factors developing acute myocardial infarction (AMI) at a relatively young age (<50-60 years old). At the other end of the spectrum, there are patients with a "full-house" CV risk factors with minor or no coronary artery disease. These suggest the presence of other factors that predispose these patients to AMI.Recent advancements in technology have led to exciting developments in our understanding of the development and prevention of CVD and AMI. The use of "big data" and "deep learning", advancements in genomics, metabolomics, and proteomics have the possibility of transforming this field. Modern prospective population-based studies aim to reclassify CV risk using integrated clinical and molecular biosignatures. However, these studies are based primarily in Western populations. Ethnic differences in CVD exist and currently in Asia, there is a dearth of such advanced data. In addition, in the Singapore Myocardial Infarction Registry (SMIR), it was reported about 1 in 4 of the AMI patients were aged 60 years or less from 2016 to 2020. The average number of AMI cases were about 900 and 2000 in patients aged < 50 years and aged between 50-59 years respectively. In term of ethnic distribution of the AMI population, about 50% of young AMI patients were Chinese, followed by Malays and Indian. In this study, the investigators specifically aim to identify novel gene variants and novel protein/metabolite candidates associated with the onset of MI in relatively young Chinese,Malay and Indian patients with minimal standard CV risk factors such as diabetes, obesity, hypertension and hypercholesterolaemia. Through these omics-based analyses, these may therefore seek to help answer some of these questions and better improve our understanding of the development of CVD and MI, potentially developing novel preventive measures to reduce the risk or delay the onset and tailoring management plans to improve treatment outcomes and reduce adverse events for the young patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult >21 years old.
2. Age ≤50 years old irrespective of the presence of CV risk factors* at the time of myocardial infarction OR Age 51-60 years old with no more than 2 CV risk factor* at the time of myocardial infarction, excluding diabetes mellitus
3. Able to provide informed consent.
4. Patients who are willing and able to comply with the study visit and procedures.
5. Prior type 1 myocardial infarction with angiographically/CT documented significant stenosis of ≥50% in LM or ≥70% in major epicardial/branch vessel (e.g. LAD, LCX, RCA).
6. Patients who are from the three main races (Chinese, Malay, Indian). Race is self-identified by patient.

   * Hypertension, hyperlipidemia, diabetes mellitus, obesity, current smoker

Exclusion Criteria:

1. Known familial hypercholesterolaemia, known vasculitides, end-stage renal disease and congenital heart disease.
2. Prior PAD and Stroke
3. Female patients who are pregnant
4. Patients who are non-Asian

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Relatively young patients with minimal cardiovascular risk factors who develop AMI from the respective public hospitals in Singapore
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
To identify novel gene variants associated with the onset of MI in relatively young patients | 5 years
  Any new genetic variants through genomic analyses

SECONDARY OUTCOMES:
To identify other novel biomarkers such as proteins, lipids and metabolites, associated with MI in young adults | 5 years
  Any new biomarkers during metabolomics and proteomics analyses

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Yap, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Participants will be assigned to a research ID, that only research coordinators and team knows

REFERENCES:
- [Background] Alwan A, Maclean DR, Riley LM, d'Espaignet ET, Mathers CD, Stevens GA, Bettcher D. Monitoring and surveillance of chronic non-communicable diseases: progress and capacity in high-burden countries. Lancet. 2010 Nov 27;376(9755):1861-8. doi: 10.1016/S0140-6736(10)61853-3. Epub 2010 Nov 10. PMID 21074258
- [Background] Shah SH, Granger CB, Hauser ER, Kraus WE, Sun JL, Pieper K, Nelson CL, Delong ER, Califf RM, Newby LK; MURDOCK Horizon 1 Cardiovascular Disease Investigators. Reclassification of cardiovascular risk using integrated clinical and molecular biosignatures: Design of and rationale for the Measurement to Understand the Reclassification of Disease of Cabarrus and Kannapolis (MURDOCK) Horizon 1 Cardiovascular Disease Study. Am Heart J. 2010 Sep;160(3):371-379.e2. doi: 10.1016/j.ahj.2010.06.051. PMID 20826242
- [Background] Bild DE, Detrano R, Peterson D, Guerci A, Liu K, Shahar E, Ouyang P, Jackson S, Saad MF. Ethnic differences in coronary calcification: the Multi-Ethnic Study of Atherosclerosis (MESA). Circulation. 2005 Mar 15;111(10):1313-20. doi: 10.1161/01.CIR.0000157730.94423.4B. PMID 15769774
- [Background] Clarke R, Peden JF, Hopewell JC, Kyriakou T, Goel A, Heath SC, Parish S, Barlera S, Franzosi MG, Rust S, Bennett D, Silveira A, Malarstig A, Green FR, Lathrop M, Gigante B, Leander K, de Faire U, Seedorf U, Hamsten A, Collins R, Watkins H, Farrall M; PROCARDIS Consortium. Genetic variants associated with Lp(a) lipoprotein level and coronary disease. N Engl J Med. 2009 Dec 24;361(26):2518-28. doi: 10.1056/NEJMoa0902604. PMID 20032323
- [Background] Wang F, Xu CQ, He Q, Cai JP, Li XC, Wang D, Xiong X, Liao YH, Zeng QT, Yang YZ, Cheng X, Li C, Yang R, Wang CC, Wu G, Lu QL, Bai Y, Huang YF, Yin D, Yang Q, Wang XJ, Dai DP, Zhang RF, Wan J, Ren JH, Li SS, Zhao YY, Fu FF, Huang Y, Li QX, Shi SW, Lin N, Pan ZW, Li Y, Yu B, Wu YX, Ke YH, Lei J, Wang N, Luo CY, Ji LY, Gao LJ, Li L, Liu H, Huang EW, Cui J, Jia N, Ren X, Li H, Ke T, Zhang XQ, Liu JY, Liu MG, Xia H, Yang B, Shi LS, Xia YL, Tu X, Wang QK. Genome-wide association identifies a susceptibility locus for coronary artery disease in the Chinese Han population. Nat Genet. 2011 Mar 6;43(4):345-9. doi: 10.1038/ng.783. PMID 21378986
- [Background] Ozaki K, Ohnishi Y, Iida A, Sekine A, Yamada R, Tsunoda T, Sato H, Sato H, Hori M, Nakamura Y, Tanaka T. Functional SNPs in the lymphotoxin-alpha gene that are associated with susceptibility to myocardial infarction. Nat Genet. 2002 Dec;32(4):650-4. doi: 10.1038/ng1047. Epub 2002 Nov 11. PMID 12426569